CLINICAL TRIAL: NCT02250898
Title: Massage for Pain and Mobility in Post-Breast Surgery Patients
Brief Title: Massage for Post Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Ash Sehgal, Director, Center for Reducing Health Disparities, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB13-01052
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Postmastectomy Lymphedema Syndrome; Pain; Shoulder Mobility Impairment; Breast Surgery
Keywords: Post Breast Surgery; Myofascial Massage; Pain; Mobility Limitations
MeSH Terms: conditions — Pain; Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental/Myofascial (Experimental): The intervention group will receive Myofascial Massage Therapy specific to breast/chest/shoulder of the affected side(s). These massages will include a variety of techniques specifically aimed at reducing pain, inflammation, and tissue sensitivity while also increasing mobility by breaking up scar tissue and thick fibrosis. The intervention massages will include the following specific techniques: skin glide, j stroking, vertical stroking, strumming, fascial stretch, circular friction, deep fascial restriction release, arm pull, side latissimus dorsi stretch, twisting, moist heat application, cold therapy, and lymphatic drainage. These massages will be twice a week at 30 minutes per massage for a period of 2 months after study enrollment.
  Interventions: Other: Myofascial Massage Therapy
- Control/Global Relaxation (Active Comparator): The control group will receive a general full body massage referred to as a Global Relaxation massage. The massage technique used here will be relaxation massage, avoiding the breast/chest/arm area. This includes light kneading and stroking in order to restore a sense of well- being. The relaxation massage will also be twice a week at 30 minutes per massage for a period of 2 months, avoiding the area of the affected shoulder/shoulders. In this way they are still being seen and touched by a massage therapist, without receiving the intervention treatment.
  Interventions: Other: Global Relaxation Massage

INTERVENTIONS:
Other: Myofascial Massage Therapy — Myofascial Massage Therapy is a manual massage therapy consisting of the following techniques: fascial stretch, circular friction, deep fascial restriction release, arm pull, side latissimus dorsi stretch, twisting, moist heat application, cold therapy, and lymphatic drainage.
  Arms: Experimental/Myofascial
Other: Global Relaxation Massage — Global Relaxation Massage is a manual massage therapy consisting of a full body relaxation massage that includes light kneading and stroking in order to restore a sense of well- being
  Arms: Control/Global Relaxation

SUMMARY:
The aims of this study are to determine the effectiveness of myofascial massage specific to the breast/chest/shoulder area in reducing self-reported pain and increasing mobility among patients who have undergone a mastectomy or other breast surgery compared to a control group receiving global relaxation massages.

DETAILED DESCRIPTION:
Post-operative breast surgery patients may face an array of complications. Breast surgery can include biopsy, lumpectomy, mastectomy or some type of reconstruction (Drackley 2012). Chronic pain and lack of mobility in the chest and/or shoulder are two of the more common and persistent issues in this population, however it is still unclear as to how many actually suffer from these (Wallace 1996). Current treatment for each of these usually includes prescribed narcotic pain medication and/or some physical therapy, the first being a treatment with many side effects, the latter being quite expensive. Global and integrated massage techniques have been used as a way of decreasing stress, anxiety, and some self-reported pain, however a targeted massage technique geared towards the breast/chest/shoulder region has not been rigorously evaluated (Drackley 2012). Myofascial massage has been shown to be an effective treatment for other post-surgical patients in reducing pain and increasing mobility, but efficacy has yet to be shown specifically in post-breast surgery patients (FitzGerald 2009). If proven effective, myofascial massage could be used as an inexpensive and non-invasive addition to current pain and mobility treatment (Cassileth 2004).

Specific Aims

Aim A.

Determine the effectiveness of myofascial massage specific to the breast/chest/shoulder area in reducing self-reported pain among patients who have undergone a mastectomy or other breast surgery.

Aim B.

Determine the effectiveness of myofascial massage specific to the breast/chest/shoulder area in increasing self-reported mobility in the affected shoulder among patients who have undergone a mastectomy or other breast surgery.

Hypothesis: Compared to control patients receiving general full body massage, myofascial massage specific to the breast/chest/shoulder area reduces pain and increases mobility in patients who have undergone breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age range 21-79 years of age
* Female
* Breast and/or axillary surgery
* 2-18 months post-operative
* Meets minimum pain and/or lack of mobility threshold as determined by survey
* Ability to give informed consent
* Ability to complete adherence task
* Benign or malignant forms of disease

Exclusion Criteria:

* History of blood clots
* Mentally incompetent
* Non-English speaking
* Infected sites or open wounds
* Currently lactating
* Currently receiving massage therapy for breast surgery
* Currently taking anticoagulants including:

Cilostazol Clopidogrel Ticlopidine Prasugrel Ticagrelor Dipyridamole Warfarin Dabigatran Rivaroxaban Apixaban Abciximab Eptifibatide Tirofiban Dalteparin Enoxaparin Fondaparinux Heparin Tinzaparin Argatroban Bivalirudin Lepirudin

Ages: 21 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in self reported pain pre and post study | 2 months
  Self report survey of current pain type and intensity will be given at the beginning of enrollment and then again after the 2 month study period ends. Pain scores will be measured pre and post.

SECONDARY OUTCOMES:
Change in self reported mobility pre and post study | 2 months
  Self report survey of current mobility issues and restrictions in relation to the breast/chest/shoulder area will be given at the time of enrollment and after the 2 month study period.

CONTACTS AND LOCATIONS:
Overall Officials: Ashwini Sehgal, MD, Principal Investigator — Ctr for Reducing Health Disparities
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Cassileth BR, Vickers AJ. Massage therapy for symptom control: outcome study at a major cancer center. J Pain Symptom Manage. 2004 Sep;28(3):244-9. doi: 10.1016/j.jpainsymman.2003.12.016. PMID 15336336
- [Background] Drackley NL, Degnim AC, Jakub JW, Cutshall SM, Thomley BS, Brodt JK, Vanderlei LK, Case JK, Bungum LD, Cha SS, Bauer BA, Boughey JC. Effect of massage therapy for postsurgical mastectomy recipients. Clin J Oncol Nurs. 2012 Apr;16(2):121-4. doi: 10.1188/12.CJON.121-124. PMID 22459520
- [Background] Fernandez-Lao C, Cantarero-Villanueva I, Diaz-Rodriguez L, Fernandez-de-las-Penas C, Sanchez-Salado C, Arroyo-Morales M. The influence of patient attitude toward massage on pressure pain sensitivity and immune system after application of myofascial release in breast cancer survivors: a randomized, controlled crossover study. J Manipulative Physiol Ther. 2012 Feb;35(2):94-100. doi: 10.1016/j.jmpt.2011.09.011. Epub 2011 Oct 21. PMID 22018755
- [Background] FitzGerald MP, Anderson RU, Potts J, Payne CK, Peters KM, Clemens JQ, Kotarinos R, Fraser L, Cosby A, Fortman C, Neville C, Badillo S, Odabachian L, Sanfield A, O'Dougherty B, Halle-Podell R, Cen L, Chuai S, Landis JR, Mickelberg K, Barrell T, Kusek JW, Nyberg LM; Urological Pelvic Pain Collaborative Research Network. Randomized multicenter feasibility trial of myofascial physical therapy for the treatment of urological chronic pelvic pain syndromes. J Urol. 2009 Aug;182(2):570-80. doi: 10.1016/j.juro.2009.04.022. Epub 2009 Jun 17. PMID 19535099
- [Background] Khan SA, Apkarian AV. The characteristics of cyclical and non-cyclical mastalgia: a prospective study using a modified McGill Pain Questionnaire. Breast Cancer Res Treat. 2002 Sep;75(2):147-57. doi: 10.1023/a:1019685829799. PMID 12243507
- [Background] Martin ML, Hernandez MA, Avendano C, Rodriguez F, Martinez H. Manual lymphatic drainage therapy in patients with breast cancer related lymphoedema. BMC Cancer. 2011 Mar 9;11:94. doi: 10.1186/1471-2407-11-94. PMID 21392372
- [Background] Wallace MS, Wallace AM, Lee J, Dobke MK. Pain after breast surgery: a survey of 282 women. Pain. 1996 Aug;66(2-3):195-205. doi: 10.1016/0304-3959(96)03064-3. PMID 8880841